CLINICAL TRIAL: NCT06760000
Title: Establishment of a Multicenter Longitudinal Cohort of Sleep With Long-term Monitoring at Home
Brief Title: S365: A Multicenter Longitudinal Cohort of Sleep Health
Acronym: S365
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Leng Yue, Associate Professor, Peking University
Other Study IDs: IRB00001052-23207
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Sleep Disorder; Sleep
Keywords: Sleep Disorder; Home Monitoring; Multicenter Longitudinal Cohort
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Five seasons Sleep Tracking Mat — Non-contact mat monitoring sleep data through pulse wave detection

SUMMARY:
The goal of this observational study is to explore the long-term health outcomes of sleep disorders in adults aged 18 and older, as well as to identify associated biomarkers and risk factors. The main questions it aims to answer are:

* What are the long-term health risks associated with sleep disorders, such as cognitive decline, cardiovascular diseases, or metabolic conditions?
* Are there specific biomarkers or patterns that can predict the onset or progression of sleep disorders?

Participants diagnosed with sleep disorders (e.g., insomnia, sleep apnea) or identified as healthy controls will undergo home-based sleep monitoring and complete clinical assessments at baseline and during follow-ups over a 3-year period. Biological samples, including blood and stool, will also be collected to analyze potential biomarkers. Data will be used to develop predictive models for sleep disorder risk and outcomes.

DETAILED DESCRIPTION:
Sleep is a vital component of overall health and well-being. However, millions of people suffer from sleep disorders, including insomnia, sleep apnea, and parasomnias, which significantly impact their quality of life and contribute to various health conditions such as cardiovascular disease, diabetes, and cognitive decline. This comprehensive observational study aims to revolutionize the understanding, diagnosis, and treatment of sleep disorders through advanced data collection, innovative technology, and cutting-edge analysis.

Study Objectives

This study focuses on building a multicenter, multidimensional clinical sample database and integrating it with big data analysis platforms to address critical gaps in sleep disorder management. Key objectives include:

1. Establishing a Standardized Database: Creating a repository of clinical, biochemical, and imaging data to better understand sleep disorders and their associated conditions.
2. Developing Predictive Models: Identifying biomarkers and risk factors to develop models for early diagnosis and risk prediction.
3. Improving Intervention Outcomes: Evaluating the long-term effects of various interventions on sleep disorders to inform personalized treatment plans.
4. Promoting Preventive Measures: Building comprehensive early warning systems for sleep disorders to prevent progression and related health issues.

Key Research Questions

* What are the biological, behavioral, and environmental factors that contribute to sleep disorders?
* How do sleep disorders progress over time, and what health risks are associated with them?
* Can specific biomarkers predict the onset or severity of sleep disorders?
* What are the long-term effects of various interventions, and how can they be optimized for individual patients?

Study Participants

This study includes two participant groups:

1. Sleep Disorder Patients: Individuals diagnosed with conditions like insomnia, sleep apnea, and parasomnia. Diagnosis is conducted through advanced techniques like polysomnography (PSG).
2. Healthy Control Group: Individuals with no reported sleep issues, serving as a comparison baseline.

Eligibility Criteria:

* Adults aged 18 or older.
* Willing to provide informed consent and participate in the study for up to three years.
* Exclusion criteria include severe mental illnesses, pregnancy, or certain medical conditions that might interfere with the study.

Study Design

This is a non-interventional cohort study designed to gather extensive, high-quality data over time. It employs both retrospective and prospective approaches to ensure comprehensive insights into sleep disorders.

1. Data Collection Methods:

   * Clinical Assessments: Participants provide demographic, lifestyle, and medical history information through standardized questionnaires.
   * Biological Samples: Blood and stool samples are collected for biochemical and microbiome analyses.
   * Sleep Monitoring: State-of-the-art technologies are used to track sleep patterns and physiological parameters.
2. Follow-Up Plan:

   * Participants are monitored at baseline and followed up annually for three years (12, 24, and 36 months).
   * Follow-ups include sleep assessments, biological sampling, and health status updates.
3. Technology Utilized:

   * Sleep Monitoring Mats: Non-contact devices placed under pillows or mattresses to measure heart rate, breathing patterns, and sleep cycles.
   * Wearable Devices: Devices like EmbracePlus and pulse oximeters continuously monitor physiological metrics, including blood oxygen levels and activity patterns.
   * Data Management Platforms: A centralized system ensures secure data storage and facilitates seamless analysis across multiple centers.

Study Outcomes

1. Primary Outcomes:

   * Identification of long-term health risks linked to sleep disorders, such as cognitive impairment, cardiovascular disease, and metabolic dysfunctions.
   * Evaluation of disease progression in participants over the study period.
2. Secondary Outcomes:

   * Discovery of biomarkers that can serve as early warning signals for sleep-related health issues.
   * Development of personalized risk models to guide early interventions.
3. Exploratory Outcomes:

   * Insights into the microbiome's role in sleep disorders through stool sample analysis.
   * Advanced imaging and EEG data to explore brain activity changes in sleep-disordered individuals.

Innovative Aspects

This study is groundbreaking in its approach:

1. Multicenter Design: Collaborates with top institutions, including Peking University and other leading hospitals, ensuring diverse and representative data.
2. Advanced Technology: Combines wearable, non-contact, and traditional monitoring devices for comprehensive data collection.
3. Big Data Integration: Leverages machine learning and advanced statistical methods to analyze high-dimensional datasets and uncover new insights.
4. Patient-Centric Approach: Ensures minimal disruption to participants' daily lives through non-invasive monitoring and easy-to-use devices.

Participant Experience

Participants play an active role in shaping the future of sleep health. Here's what they can expect:

1. Initial Visit:

   * Comprehensive clinical assessment.
   * Baseline sleep study using wearable or non-contact devices.
   * Collection of blood and stool samples.
2. Follow-Up Visits:

   * Annual updates on sleep quality and overall health through home-based monitoring.
   * Feedback sessions where participants can learn about their sleep health and contribute valuable data for scientific progress.
3. Supportive Measures:

   * Access to technical support for using monitoring devices.
   * Regular check-ins from the research team to ensure a smooth participation experience.

Benefits of Participation

Participants can benefit in several ways:

* Gain valuable insights into their sleep health and overall well-being.
* Contribute to cutting-edge research that may lead to better diagnostics and treatments.
* Help improve public health by advancing the understanding of sleep disorders and their impact on society.

Ethical Considerations

The study adheres to the highest ethical standards to ensure participant safety and data integrity:

* Informed Consent: Participants receive detailed information about the study and must provide written consent before participation.
* Data Anonymization: All data collected are de-identified to protect participants' privacy.
* Ethical Oversight: The study is approved and monitored by the Peking University Biomedical Ethics Committee, ensuring compliance with ethical guidelines.

Collaborating Institutions

This research is a collaborative effort led by Peking University, involving:

* Sichuan University: Focus on chronic insomnia and narcolepsy.
* Shanghai Jiao Tong University: Expertise in sleep apnea.
* Central South University: Research on parasomnia and other sleep disorders.
* Additional Regional Centers: Providing diverse patient data and technical support.

Long-Term Vision

The study aims to create a lasting impact:

1. Transforming Diagnosis and Treatment: Establishing evidence-based guidelines for early detection and effective interventions.
2. Empowering Health Care Providers: Providing tools and resources to enhance clinical practice.
3. Educating the Public: Raising awareness about the importance of sleep health and its impact on overall well-being.

How Families and Health Care Providers Can Help

Families and health care providers are integral to the study's success:

* Support Participants: Encourage adherence to monitoring and follow-up schedules.
* Promote Awareness: Help participants recognize the importance of sleep health.
* Collaborate with Researchers: Provide feedback and share observations to enrich the study's findings.

Call to Action

This study offers an unprecedented opportunity to advance sleep science and improve millions of lives. By participating or supporting the research, individuals and health care providers can contribute to a brighter, healthier future for those affected by sleep disorders. Let's work together to unlock the mysteries of sleep and transform care for generations to come.

ELIGIBILITY:
Inclusion Criteria:

* Willing to voluntarily participate in the study and provide signed informed consent.
* Gender is not restricted, and baseline age is 18 years or older.
* Experiencing sleep disorders and capable of complying with the study procedures and tests.

Exclusion Criteria:

* Diagnosed with severe mental health conditions, such as bipolar disorder, schizophrenia, or claustrophobia.
* Suffering from infectious diseases, including tuberculosis, HIV/AIDS, or syphilis.
* Pregnant women.
* Experiencing acute inflammatory responses at the time of enrollment.
* Long-term use of corticosteroids or undergoing hormone replacement therapy.
* Determined by the researcher to be unsuitable for participation for any reason.
* Patients with specific diseases (e.g., cardiovascular conditions) may be excluded if the study focuses on related comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include adults aged 18 years and older, recruited from two primary sources: clinical sleep centers and online advertisements. Participants will be divided into two groups: those diagnosed with sleep disorders, including insomnia, sleep apnea, and parasomnia, and healthy controls with no clinical symptoms. Individuals with sleep disorders will be identified through polysomnography or equivalent diagnostic methods, ensuring accurate categorization.
  Recruitment will target a diverse population to reflect a broad range of demographic and lifestyle factors, such as age, gender, and socio-economic background. The healthy control group will include individuals diagnosed as free from sleep-related conditions during clinical evaluations or through self-reported health statuses verified by researchers.
  Exclusion criteria include individuals with severe mental illnesses (e.g., bipolar disorder, schizophrenia), infectious diseases (e.g., tuberculosis, HIV/AIDS), pregnan
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Sleep Disorders and Related Diseases | 36 months (Baseline and follow-ups at 12, 24, and 36 months)
  * Measure the occurrence of sleep disorders and related diseases, including cognitive decline, cardiovascular diseases, and metabolic conditions, over the follow-up period.
  * Data will be collected through clinical evaluations, sleep monitoring (e.g., polysomnography, wearable devices), and laboratory analyses (e.g., blood biomarkers).
  * Key metrics include the development or progression of these conditions, assessed through standardized diagnostic criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medical Technology, Peking University Health Science Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the individual participant data (IPD) that are necessary for presenting the results included in publications. This will include de-identified data related to key outcomes, such as demographic information, clinical assessments, and sleep monitoring results. Additional data beyond what is included in the publications may be available upon reasonable request. Researchers interested in accessing these data should contact the project lead, who will evaluate requests on a case-by-case basis to ensure compliance with ethical and legal guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR